CLINICAL TRIAL: NCT06545617
Title: A Phase 1b/2, Multicenter, Open-Label Study of BAT8006, an Anti- FRα Antibody Drug Conjugate (ADC) for Platinum-resistant Ovarian Cancer Subjects
Brief Title: A Clinical Study to Observe How Well That BAT8006 Works on Patients With Platinum Resistance Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Reconsideration of the subsequent international development of BAT8006
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8006-002-CR
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Platinum-resistant Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): BAT8006 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8006 for Injection
- Cohort 2 (Active Comparator): BAT8006 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8006 for Injection
- Cohort 3 (Active Comparator): BAT8006 for Injection does according to protocol (frequency: Q3W)
  Interventions: Drug: BAT8006 for Injection

INTERVENTIONS:
Drug: BAT8006 for Injection — Intravenous infusion: once every three weeks.The infusion time in the first cycle is recommended to be ≥ 90 minutes. If no infusion reaction occurs, the subsequent cycle can be completed within 30~60 minutes.
  Other Names: Recombinant humanized anti-FRα monoclonal antibody-Exatecan conjugate

SUMMARY:
This is a Phase 1b/2, open-label, 2-part, global study designed to investigate the anti-tumor activity as well as the safety and efficacy of BAT8006 in subjects with platinum resistance ovarian cancer

DETAILED DESCRIPTION:
Part 1 is a Dose Finding Study. The RP2D will be confirmed in Part 1, and this RP2D will be further evaluated in Part 2. In Part 1, PK samples will be collected and analyzed to support the determination of RP2D. Three dose cohorts are planned. Subjects will be assigned to these three dosages in parallel.

Part 2 will expose subjects at the RP2D confirmed in Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give voluntary informed consent and understand the study and are willing to follow and complete all the study required procedures.
2. Women ≥ 18 years old.
3. Subjects with histologically or cytologically confirmed platinum-resistant, advanced or metastatic epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer.
4. Presence of at least one measurable lesion per RECIST v1.1. that was not in a prior radiation or other locally treated area.
5. Life expectancy ≥ 3 months.
6. Adequate hematological, liver, kidney and coagulation function.

Exclusion Criteria

1. Females who are pregnant or nursing.
2. Had major surgery within 28 days of the Screening visit.
3. History of autologous transplantation ≤ 3 months
4. History of severe infection deemed clinically significant by the PI or designee within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose of study drug.
5. History of human immunodeficiency virus (HIV) infection.
6. Active hepatitis B or C.
7. Any other serious underlying medical.
8. Received cancer-directed therapy within the timeframes.
9. Subjects have other active malignancies within 5 years prior to the first dose.
10. Known allergies, hypersensitivity, or intolerance to the study drug or its excipients.
11. Vaccinated with any live-attenuated vaccine within 4 weeks.
12. Subjects with known history of psychiatric disorders, drug abuse, alcoholism or drug addiction.
13. Subjects who are estimated by the investigator to have poor compliance with the clinical study or who have other factors that are not appropriate to participate in the study in the opinion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) and/or identify the recommended Phase 2 dose (RP2D) of BAT8006 | At the end of Cycle 1 (each cycle is 21 days)
  Incidence of dose-limiting toxicities (DLTs)
The tolerability of BAT8006 | From date of first dose administration until the date of clinical progression, adverse event, physician decisionor or date of death from any cause, whichever came first, assessed at most up to 27 months
  Frequency and duration of dose interruptions and reductions
Adverse events（AE） | From signed ICF to 30 days after the last drug administration
  Include SAEs, TEAEs
Physical examination | From signed ICF to 30 days after the last drug administration
  Number of participants with abnormal physical examination findings
ECOG | From signed ICF to 30 days after the last drug administration
  Changes in ECOG score
Vital signs | From signed ICF to 30 days after the last drug administration
  Number of participants with abnormal vital signs
Laboratory testings | From signed ICF to 30 days after the last drug administration
  Number of participants with abnormal laboratory testing results
Electrocardiogram（ ECG ） | From signed ICF to 30 days after the last drug administration
  Number of participants with abnormal ECG results
Echo/MUGA | From signed ICF to 30 days after the last drug administration
  Number of participants with abnormal Echo/MUGA results
Ophthalmologic findings | From signed ICF to 30 days after the last drug administration
  Number of participants with abnormal ophthalmologic findings

SECONDARY OUTCOMES:
The immunogenicity of BAT8006 | Pre-dose of Cycle 1 to Cycle 1 Day 15, Pre-dose of Cycle 2, 4 until every 4 cycles
  Specification and quantification of ADAs or NAb
Objective response rate (ORR) | From signed ICF to 30 days after the last drug administration
  The proportion of subjects who achieved a confirmed response of complete response (CR) or partial response [PR]
Duration of response (DOR) | From signed ICF to 30 days after the last drug administration
  The time between the first assessment of objective remission of a tumor and death from any cause before the first assessment of Disease progression (PD)
Best percent change in the sum of the longest diameters (SLD) of measurable tumors | From signed ICF to 30 days after the last drug administration
  Best percent change in the sum of the longest diameters (SLD) of measurable tumors according to RECIST v1.1
Progression-free survival (PFS) | From signed ICF to 30 days after the last drug administration
  The time from the date of randomization/registration to the earlier of the dates of the first objective documentation of radiographic PD via independent radiologic facility review based on RECIST version 1.1 or death due to any cause
The pharmacokinetics (PK) profile of BAT8006（Maximum concentration (Cmax)） | Cycle 1 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 2 Day 1; Cycle 3 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 4/6/8/12/16/20/24/28/32 Day 1
  Maximum concentration (Cmax)
The pharmacokinetics (PK) profile of BAT8006（Time of Cmax (Tmax)） | Cycle 1 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 2 Day 1; Cycle 3 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 4/6/8/12/16/20/24/28/32 Day 1
  Time of Cmax (Tmax)
The pharmacokinetics (PK) profile of BAT8006（Area under the curve (AUC)） | Cycle 1 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 2 Day 1; Cycle 3 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 4/6/8/12/16/20/24/28/32 Day 1
  Area under the curve (AUC)
The pharmacokinetics (PK) profile of BAT8006（Terminal half-life (t½)） | Cycle 1 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 2 Day 1; Cycle 3 Day 1, 2, 3, 4, 8, 15, 22 to Cycle 4/6/8/12/16/20/24/28/32 Day 1
  Terminal half-life (t½)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, Principal Investigator — The University of Oklahoma College of Medicine